CLINICAL TRIAL: NCT06650150
Title: Comparative Study on Respiratory Muscle Strength and Exercise Capacity in Smokers With COPD, PRISm and Pre-COPD
Brief Title: Respiratory Muscle Strength and Exercise Capacity in Smokers
Acronym: mip
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Sabri Serhan OLCAY, Assistant Professor, Muğla Sıtkı Koçman University
Other Study IDs: MIP24
Record Dates: First submitted 2024-10-11; First posted 2024-10-21 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: COPD - Chronic Obstructive Pulmonary Disease
Keywords: PRISm; Pre-COPD; COPD; MIP; 6mwt
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Maximal Respiratory Pressures; Walk Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- PRISm: cigarette smokers with FEV1 below 80%
  Interventions: Diagnostic Test: maximal inspiratory pressure; Diagnostic Test: maximal expiratory pressure; Diagnostic Test: 6 minute walk test
- preCOPD: cigarette smokers with normal pft
  Interventions: Diagnostic Test: maximal inspiratory pressure; Diagnostic Test: maximal expiratory pressure; Diagnostic Test: 6 minute walk test
- COPD: cigarette smokers with FEV1/FVC less than 70%
  Interventions: Diagnostic Test: maximal inspiratory pressure; Diagnostic Test: maximal expiratory pressure; Diagnostic Test: 6 minute walk test

INTERVENTIONS:
Diagnostic Test: maximal inspiratory pressure — maximal inspiratory pressure (mip) will be measured with a specific device
Diagnostic Test: maximal expiratory pressure — MEP will be measured with a specific device
Diagnostic Test: 6 minute walk test — 6mwt will be done by a phsyotherapist

SUMMARY:
This cross-sectional study aims to evaluate the respiratory muscle strength and physical capacity of symptomatic adult smokers in Muğla. The study population will be the patients who were admitted to the pulmonary outpatient clinic of Muğla Training and Research Hospital between July 2024 and December 2024. The primary outcome is the proportion of individuals with Maximum Inspiratory Pressure (MIP) below 80%. Secondary outcomes include the 6-Minute Walk Test (6MWT) distance, Maximum Expiratory Pressure (MEP), and COPD Assessment Test (CAT) scores. Smokers will be categorized into COPD, PRISm, and Pre-COPD groups. The study will adjust for BMI as a key confounder and assess the modifying effects of gender, smoking habits, and age. Ethical approval and informed consent will be obtained, with data analysis focusing on descriptive statistics, comparative analysis, and regression models to understand the impact of smoking on respiratory health.

ELIGIBILITY:
Inclusion Criteria:

* At least 5 packages of cigarette smokers who have an appropriate PFT done at our lab. (pulmonary function test must be performed at evaluable standards according to ERS/ATS guidelines)

Exclusion Criteria:

* Respiratory infection at the time of measurement (upper or lower resp. tract, viral or bacterial infections)
* Presence of chronic respiratory diseases (Asthma, IPF, Bronchiectasis, [except COPD])
* Exacerbation due to chronic respiratory diseases (except mild COPD exacerbation)
* Neuromuscular disease (ALS, Guillain-Bare syndrome, Muscular dystrophies, Myasthenia gravis)
* Restrictive pulmonary disease (IPF, Sarcoidozis, Progresif Pulmonary Fibrosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of symptomatic smokers admitted to the pulmonary outpatient clinic of Muğla Training and Research Hospital between July 2024 and December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-10-20 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
MIP | day 1
  MIP<80% in each grous

SECONDARY OUTCOMES:
MEP | day 1
  mep< 80% in each group

OTHER OUTCOMES:
6MWT | day 1
  6MWT distance in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Muğla Training and Research Hospital, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided